CLINICAL TRIAL: NCT06426368
Title: " Prognostic Value of Soluble ST2 Beyond B-Type Natriuretic Peptide in Management of Patients With Heart Failure"
Brief Title: Soluble ST2 in Patients With Heart Failure"
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed Hesham Ahmed Mohamed, doctor, Assiut University
Other Study IDs: ST2 in H.F patients
Record Dates: First submitted 2024-05-12; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: HF with reduced ejection fraction (HFrEF, LVEF ≤ 40%)
  Interventions: Diagnostic Test: ST2
- Group II: HF with mildly reduced ejection fraction (HFmrEF, LVEF 41-49%)
  Interventions: Diagnostic Test: ST2
- Group III: HF with preserved ejection fraction (HFpEF, LVEF ≥ 50%)
  Interventions: Diagnostic Test: ST2

INTERVENTIONS:
Diagnostic Test: ST2 — ELISA used to detect levels of ST2 and BNP as inflammatory biomarkers in patients with heart failure
  Other Names: BNP

SUMMARY:
1. The aim of this study was to explore the relationship between peripheral circulating serum soluble suppression of tumorigenicity-2 (sST2) levels and inflammatory biomarkers in patients with heart failure
2. Additive role of sST2 to NPs in of heart failure patients

DETAILED DESCRIPTION:
Heart failure (HF), a complex and heterogeneous medical syndrome characterized by structural and functional cardiac abnormalities and hemodynamic disruptions, represents the end-stage manifestation of numerous cardiovascular disorders . HF is categorized into three groups based on the measurement of the left ventricular (LV) ejection fraction (LVEF) according to the European Society of Cardiology (ESC) Guidelines issued in 2021: HF with reduced ejection fraction (HFrEF, LVEF ≤ 40%), HF with mildly reduced ejection fraction (HFmrEF, LVEF 41-49%), and HF with preserved ejection fraction (HFpEF, LVEF ≥ 50%) .

Quantifying concentrations of circulating biomarkers plays a major role in most cardiovascular (CV) diseases, including (HF) .

An ideal biomarker in HF should be measured non-invasively and at low cost, highly sensitive to allow for the early detection of the disease .

N-terminal pro-B-type natriuretic peptide (NT-proBNP) released by cardiac muscle tissue in response to abnormal volume load is an established indicator for the diagnosis and prognosis of HF .

However, there are important limitations to natriuretic peptide (NP) testing in HF .

Soluble suppression of tumorigenicity-2 (sST2) is the circulating form of the interleukin-33 membrane receptor released in response to inflammation, fibrosis in various organs, and myocardium stress .

Soluble (s)ST2 has been proposed as a useful biomarker for heart failure (HF) patient management. Myocardial damage or mechanical stress stimulate sST2 release. ST2 competes with a membrane bound receptor (ST2 ligand, or ST2L) for interleukin-33 (IL-33) binding, inhibiting the effects induced by the ST2L/IL-33 interaction so that excessive sST2 may contribute to myocardial fibrosis and ventricular remodelling.

So biomarkers such as NT-proBNP and sST2 could potentially be used as surrogates for clinical outcomes in patients with HF and may be useful in monitoring disease progression and assessing the response to therapy .

ELIGIBILITY:
Inclusion Criteria:

* patients 18-80 years.
* Both sexes will be included.
* including signs and symptoms of HF (e.g., elevated jugular venous pressure and altered apical beat position), altered LVEF (< 40%; 40%-49%; ≥ 50%)

Exclusion Criteria:

* Patients <18 years
* Patients with documented evidence of cardiogenic shock .
* Patients with Acute coronary syndrome within 30 days.
* chronic kidney disease patients with glomerular filtration rate < 30
* Patients with interstitial pulmonary fibrosis .

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Chemistry unit of Clinical Pathology Department and Cardiovascular Department, Assiut University Hospitals, Assiut University, Egypt Heart failure patients will be classified according to NYHA classification
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate if Soluble ST2 is strongly associated with measures of HF severity and poor outcome | Baseline
  Study ST2 level in heart failure patients and correlate results with clinical data and other inflammatory biomarker
Evaluation of BNP and ST2 could have a potential role in prognosis. | Baseline
  Study value of BNP in prognosis and compare it with ST2

SECONDARY OUTCOMES:
• Clinical Impact and Treatment Decision Support | Baseline
  Evaluate ST2 as a novel biomarker which provide risk stratification of patients with acute and chronic HF beyond BNPs

CONTACTS AND LOCATIONS:
Overall Officials: Randa Ahmed, Study Director — Assiut University; Hanan Omer, Study Director — Assiut University; Yousra Mamdouh, Study Director — Assiut University

REFERENCES:
- [Background] Purdy GE, Payne SM. The SHI-3 iron transport island of Shigella boydii 0-1392 carries the genes for aerobactin synthesis and transport. J Bacteriol. 2001 Jul;183(14):4176-82. doi: 10.1128/JB.183.14.4176-4182.2001. PMID 11418557